CLINICAL TRIAL: NCT05986929
Title: Acceptability of a Communication Tool Using Bedside Magnetized Posters, as Well as Barriers and Facilitators to Its Use.
Brief Title: Acceptability, Barriers and Facilitators of a Communication Tool in Hospital Settings
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fondation Vitae (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-5186
Record Dates: First submitted 2023-06-30; First posted 2023-08-14 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-04

CONDITIONS: Communication, Multidisciplinary
Keywords: communication; multidisciplinary; hospital settings
MeSH Terms: conditions — Communication | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Staff on the neurology and geriatric units: Staff that will participate in the electronic survey (N=100) and focus group (N=6-8)
  Interventions: Other: focus group; Other: electronic survey

INTERVENTIONS:
Other: focus group — Two semi-structured group interviews, lasting 30-60 minutes, on facilitators and barriers to poster use by staff members (N=6-8).
Other: electronic survey — An electronic survey of 15 closed questions on the acceptability of the magnetic posters (N=100).

SUMMARY:
The presence of appropriate systems to promote good communication within the care team is one of the ten important characteristics identified for effective interdisciplinary work. However, the current communication systems at the Eastern Townships University Health and Social Services Centre of the Sherbrooke University Hospital (SUH), an hospital setting in Sherbrooke (Quebec, Canada), are numerous, scattered and difficult to identify quickly. The bedside magnetized posters were developed to address this issue. The use of this kind of tool should improve teamwork, communication, and patient care. As the bedside magnetized posters are now well established on the stroke and geriatric units at the SUH, it is essential to evaluate their acceptability by staff members. In addition, identifying the barriers and facilitators to their use will support the team for eventual deployment in other care environments at the SUH.

DETAILED DESCRIPTION:
The objectives of the study are:

1. To describe the acceptability of magnetic posters by staff members in the Neurology Department - Stroke Unit, where they are already well established, and in the Geriatric Department, where they are newly introduced.
2. To identify barriers and facilitators to the use of magnetic posters to assist the team in an eventual deployment in other care environments at SUH.

Methods

A mixed sequential design will be used (quantitative, qualitative and observational). The study population will be staff working with inpatients in the neurology-stroke and geriatric units of SUH. Staff meeting the eligibility criteria will be invited to complete an electronic survey on the acceptability of the magnetic posters. The survey will consist of 15 closed questions relating to the use of the magnetic posters (e.g. frequency of poster consultation) and its acceptability (e.g. ease of use, poster content), one open question to gather suggestions for improving the tool and 6 socio-demographic questions. The survey will take approximately 10-15 minutes to complete, and responses will be recorded on the Research Centre on Aging's RedCap server for later analysis.

Also, a member of the research team will carry out observations on the neurology-stroke and geriatric units for one half-day, in order to collect data concerning, among other things, how the posters are used (e.g. where are the posters available to staff, which posters are used) and the characteristics of the patients for whom the posters are used.

Finally, two semi-structured group interviews, one for the neurology-stroke unit and one for the geriatric unit, will be facilitated by a member of the research team. Each group will be made up of 6 to 8 employees from a variety of professions, in order to be representative of the population under study and will last 30-60 minutes. The focus groups will address the facilitators and barriers to poster use for each respective unit. Discussions will be recorded and verbatims will be kept for later analysis.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 and over
* employed by the SUH and working on stroke and geriatric units

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of staff members working with people hospitalized in the neurology-stroke and geriatric units of SUH. The sample will be made up of various types of professionals such as nurses, beneficiary attendants, physicians, residents, physiotherapists, occupational therapists, speech therapists, nutritionists, social workers, as well as people assigned to housekeeping and user transportation. If student nurses are present on these units at the time of recruitment, they may also be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Acceptability | From the time the participants begin the electronic survey to the time their answers are sent off (approx. 15 to 20 minutes). There are no cut-off points for this outcome
  questions on acceptability of the magnetic posters will be asked in the electronic survey
Barriers and facilitators | This outcome will be measured during the participants' focus group, which should have a duration of approx. 60 minutes. There are no cut-off points for this outcome
  questions on barriers and facilitators to poster use will be asked during the focus group

SECONDARY OUTCOMES:
Questionnaire on the use of the magnetic posters | This outcome will be measured during the observational half-day, which should have a duration of approx. 4 hours. There are no cut-off points for this outcome
  during the observational half-day, how the posters are used (where they are used and which posters are used) in the stroke and geriatric units will be collected
Characteristics of the patients | This outcome will be measured during the observational half-day, which should have a duration of approx. 4 hours. There are no cut-off points for this outcome
  This outcome will be measured during the observational half-day, which should have a duration of approx. 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Helene Milot, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- CIUSSS de l'Estrie CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No